CLINICAL TRIAL: NCT01558011
Title: Using Genetic Polymorphisms of Drug Metabolism and Immunohistochemical Stain to Predict the Efficacy and Toxicity in Patients With Gastric Adenocarcinoma - A Phase II Study
Brief Title: Using Genetic Polymorphisms to Predict the Efficacy and Toxicity - A Gastric Adenocarcinoma Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The budget issues.
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Tri-Service General Hospital (Other); Mackay Memorial Hospital (Other); National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T3211; 100CT202 (Other Grant/Funding Number: NRPB)
Record Dates: First submitted 2012-03-05; First posted 2012-03-20 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2013-10

CONDITIONS: Gastric Adenocarcinoma
Keywords: gastric adenocarcinoma; Capecitabine and oxaliplatin (XELOX); Docetaxel and capecitabine (TX); Using genetic polymorphisms; drug metabolism and immunohistochemical stain; predict the efficacy
MeSH Terms: interventions — Capecitabine; Oxaliplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chemotherapy (Experimental): Chemotherapy:
  Drug: Capecitabine, Oxaliplatin, Docetaxel Dosing Regimena: total of 6 cycles of modified XELOX regimen repeats every 2 weeks, and followed by 4 cycles of TX repeats every 3 weeks. After 10 cycles of treatment, patients may continue to treat with either of the regimen, preferably the one having the best efficacy.
  Interventions: Drug: Capecitabine, Oxaliplatin, Docetaxel

INTERVENTIONS:
Drug: Capecitabine, Oxaliplatin, Docetaxel — Capecitabine: 500 mg film coated tablets; Oxaliplatin: 50 mg/ 10 ml; Docetaxel: 20 mg / 0.5ml vial.
  Dosing Regimena: total of 6 cycles of modified XELOX regimen repeats every 2 weeks, and followed by 4 cycles of TX repeats every 3 weeks. After 10 cycles of treatment, patients may continue to treat with either of the regimen, preferably the one having the best efficacy.
  Other Names: Capecitabine (Xeloda○R), company: Roche; Oxaliplatin (Eloxatin○R, company: Sanofi-Avantis; Docetaxel (Taxotere○R, company: Sanofi-Avantis

SUMMARY:
This is an open-label, non-comparative phase II study of sequential capecitabine plus oxaliplatin followed by docetaxel plus capecitabine in patients with unresectable gastric adenocarcinoma.

DETAILED DESCRIPTION:
There are two primary objectives in different steps. In the first step, the primary objective of this study is to investigate the objective response rate in patients receiving sequential capecitabine plus oxaliplatin followed by docetaxel plus capecitabine in patients with unresectable gastric adenocarcinoma.

In the second step, the primary objective of this study is to screen the predictive biomarkers of three different chemotherapeutic drugs and also investigate the objective response rate in patients receiving sequential capecitabine plus oxaliplatin followed by docetaxel plus capecitabine in patients with unresectable gastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed gastric adenocarcinoma.
* At least one measurable lesion in a non-irradiated area.
* No prior exposure to systemic chemotherapy for advanced gastric cancer.
* For those have adjuvant chemotherapy after a curative gastrectomy, the last dosing of previous adjuvant chemotherapy should be at least 6 months before the start of this treatment.
* Age > 20 years old.
* ECOG Performance Status 2.
* Life expectancy greater than 12 weeks.
* Adequate bone marrow function :absolutely neutrophil count 1.5 x 109/L or WBC 4 x 109/L; Hemoglobin > 9 g/dl;platelet count 100 x 109/L.
* Adequate liver function : ALT & AST 2.5 x ULN if without liver metastasis or 5 x ULN if with hepatic metastasis. Alkaline phosphatase 2.5 x ULN if without liver metastasis or 5 x ULN, if with hepatic and bone metastasis. Bilirubin < 2 x ULN
* Adequate renal function :Creatinine < 1.5 x ULN.
* Patients must be accessible for treatment and follow-up in the participating centers.

Exclusion Criteria:

* Patient who are receiving concurrent radiotherapy, chemotherapy or other experimental therapy.(Previous radiotherapy is allowable if the last dose was given more than 2 weeks before the protocol treatment).
* Major surgery within two weeks prior to entering the study.
* Patients with CNS metastasis, including clinical suspicion.
* Patients who are under active or uncontrolled infections.
* Patients who had cardiac arrhythmia or myocardial infarction history 6 months before entry.
* Patients with clinically detectable peripheral neuropathy > 2 on the CTC criteria
* Patients with concomitant illness that might be aggravated by chemotherapy.
* Patients who are pregnant or with breast feeding.
* Other concomitant or previously malignancy within 5 yrs except for in situ cervix cancer or squamous cell carcinoma of the skin treated by surgery only.
* Patients with hypersensitivity to any component of the chemotherapeutic regimen.
* Mental status is not fit for clinical trial
* Can not take study medication orally

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Every 6 weeks
  Tumor responses in measurable lesions are to be evaluated by the tumor response guidelines validated by the Response Evaluation Criteria in Solid Tumors (RECIST) Group . The new version 1.1 was published in 2009.

SECONDARY OUTCOMES:
Progression-free survival | Every 6 weeks
  Be calculated as the duration between the first date of randomization and the date of disease recurrence or progression according to RECIST (failed), taking the status of tumor at the treatment has been completed as the reference, or death (failed), or the date of withdrawal (last contact date, censored), or the scheduled data analysis date (censored).

CONTACTS AND LOCATIONS:
Locations (1):
- National Health Research Institutes, Zhunan, Miaoli, Taiwan